CLINICAL TRIAL: NCT07288736
Title: The Distinctive Effects of Aroma-Formulas on Sundown Syndrome, Mood and Sleep Quality of Patients With Dementia
Brief Title: Aromatherapy Formulas for Sundowning and Sleep Quality in Patients With Dementia.
Acronym: AROMA-SUN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NCKU HREC-F-111-613-2
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Dementia; Sundowning
Keywords: Aromatherapy; Essential Oils; Sundowning; Sundown Syndrome; Sleep Quality; Dementia
MeSH Terms: conditions — Dementia; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Single-group, two-period crossover trial without randomization. All participants first receive Aromatherapy Formula A in Phase 1 for 2 weeks (5 days per week, twice daily diffusion at 9:00 a.m. and 2:00 p.m.), followed by a 2-week washout period. In Phase 2, the same participants receive Aromatherapy Formula B for 2 weeks with the same schedule. Each participant serves as his or her own control to evaluate changes in sundown syndrome and sleep quality.
Masking Description: This is an open-label study; no masking procedures will be used. Participants, care providers, and investigators are aware of the aroma formula administered in each treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Aromatherapy - Formula A then Formula B (Experimental): Participants will receive a two-phase aromatherapy intervention. In Phase 1, they will receive Aromatherapy Formula A for 2 weeks, followed by a 2-week washout period. In Phase 2, they will receive Aromatherapy Formula B for another 2 weeks. Aromatherapy will be administered by diffusion twice daily (09:00 and 14:00), 5 days per week, in the dementia care unit.
  Interventions: Other: Aromatherapy Formula A; Other: Aromatherapy Formula B

INTERVENTIONS:
Other: Aromatherapy Formula A — Participants receive Aromatherapy Formula A for 2 weeks. In the morning, Formula A1 (a 2:1 blend of organic rosemary and organic lemon essential oils) is diffused in the dementia care unit; in the afternoon, Formula A2 (a 2:1 blend of organic lavender and organic sweet orange essential oils) is diffused. Aromatherapy is administered by diffusion twice daily (around 09:00 and 14:00), 5 days per week, during the 2-week intervention period.
Other: Aromatherapy Formula B — Participants receive Aromatherapy Formula B for 2 weeks. Formula B is a calming compound essential oil blend containing organic sweet orange (Citrus sinensis), spike lavender (Lavandula latifolia), true lavender (Lavandula angustifolia), vetiver (Vetiveria zizanoides), bergamot (Citrus bergamia), and Roman chamomile (Chamaemelum nobile). The blend is diffused in the dementia care unit twice daily (around 09:00 and 14:00), 5 days per week, during the 2-week intervention period. In the crossover sequence, this phase follows a 2-week washout period after Formula A.

SUMMARY:
Dementia is common in aging societies and is often accompanied by sundowning syndrome and sleep problems. These symptoms can be very distressing for patients and place a heavy burden on family members and professional caregivers. Aromatherapy using essential oils, especially lavender, has shown promise in reducing behavioral symptoms in people with dementia, but evidence on compound essential oil formulas and their effects on both sundowning and sleep quality remains limited.

This study will compare two different compound essential oil formulas for people with dementia living in long-term care facilities in southern Taiwan. Each participant will receive both formulas at different times in a repeated crossover design. In Phase 1, participants will receive a stimulating formula in the morning (rosemary and lemon) and a relaxing formula in the afternoon (lavender and sweet orange). In Phase 2, they will receive a calming blend that includes sweet orange, spike lavender, true lavender, vetiver, bergamot, and Roman chamomile. Aromatherapy will be administered by diffusion twice a day, five days per week, for two weeks in each phase.

The main outcomes are changes in agitation and sleep quality, measured using the Chinese versions of the Cohen-Mansfield Agitation Inventory and the Pittsburgh Sleep Quality Index. The findings are expected to provide preliminary evidence on whether compound essential oil formulas can be a simple, non-drug approach to help manage sundowning syndrome and improve sleep in people with dementia.

DETAILED DESCRIPTION:
Dementia is increasingly prevalent in rapidly aging societies and is frequently accompanied by neuropsychiatric symptoms, including sundowning syndrome and disturbed sleep-wake cycles. Sundowning behaviors-such as agitation, wandering, and confusion that worsen in the late afternoon or evening-are particularly challenging to manage and are associated with poorer sleep quality, increased use of psychotropic medications, and heightened caregiver burden. Non-pharmacological interventions that are safe, simple, and feasible in long-term care settings are urgently needed.

Aromatherapy has emerged as a potentially useful complementary therapy for behavioral and psychological symptoms of dementia. Prior studies have suggested that lavender and other essential oils may reduce agitation and promote relaxation; however, most existing evidence focuses on single oils, small samples, or non-standardized protocols. Data on compound essential oil formulations, especially those targeting both sundowning syndrome and sleep quality, remain limited.

This study is designed to evaluate the comparative effectiveness of two compound essential oil formulas on agitation related to sundowning and on overall sleep quality in patients with dementia. A repeated crossover design will be used. Participants will be recruited from long-term care facilities in southern Taiwan and must have a medical diagnosis of dementia and observable sundowning or sleep disturbance.

The intervention includes two 2-week aromatherapy phases, separated by an appropriate washout period. Aromatherapy is delivered by diffusion in the dementia care unit twice daily (09:00 and 14:00), five days per week.

Phase 1 (Formula A):

Morning: Formula A1, a 2:1 blend of organic rosemary (Rosmarinus officinalis) and organic lemon (Citrus limon) essential oils, intended to promote alertness and daytime activity.

Afternoon: Formula A2, a 2:1 blend of organic lavender (Lavandula angustifolia) and organic sweet orange (Citrus sinensis) essential oils, intended to reduce agitation and support evening relaxation.

Phase 2 (Formula B):

Participants receive a calming compound blend (Formula B) that includes organic sweet orange, spike lavender, true lavender, vetiver, bergamot, and Roman chamomile. This formulation is designed to provide broader anxiolytic, sedative, and stabilizing effects across the day.

All essential oils are high-quality organic products, and diffusion is carried out under standardized conditions by trained staff. Usual medical and nursing care continues throughout the study.

Outcome measures focus on behavioral agitation and sleep quality. Agitation associated with sundowning is assessed using the Chinese version of the Cohen-Mansfield Agitation Inventory (CCMAI), and sleep quality is evaluated using the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI). Demographic and clinical characteristics are collected to describe the sample and to explore potential covariates.

Because each participant serves as his or her own control across the two aromatherapy sequences, data will be analyzed using a linear mixed model (LMM) to examine within-subject changes over time, while accounting for period and sequence effects. The primary comparisons will focus on differences in CCMAI and CPSQI scores between Formula A and Formula B phases.

The expected outcome is to generate preliminary clinical evidence that compound essential oil formulations can be integrated as a simple, low-risk, non-pharmacological strategy to manage sundowning symptoms and improve sleep in people with dementia. If effective, these aromatherapy protocols could be adapted for long-term care facilities, community programs, and home-based caregiving, thereby helping to reduce caregiver burden and improve quality of life for both patients and families.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia by a specialist according to DSM-5 (any type) OR SPMSQ score < 8.
* Manifesting sundown syndrome with a score ≥ 26 on the CMAI-C.
* Able to speak Mandarin or Taiwanese.

Exclusion Criteria:

* Clinical diagnosis of a psychiatric disorder (e.g., schizophrenia, bipolar disorder).
* Acute stage of illness within the past 2 weeks.
* Olfactory disorder or loss of smell (anosmia).
* Allergy to essential oil fragrances.
* Currently receiving aromatherapy.
* Respiratory disease (e.g., asthma, COPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Change in agitation/sundowning behaviors (Chinese Cohen-Mansfield Agitation Inventory, CCMAI) | Baseline and the end of each 2-week aromatherapy phase (up to 6 weeks)
  Agitation and sundowning behaviors will be assessed using the Chinese version of the Cohen-Mansfield Agitation Inventory (CCMAI). The inventory includes 29 items rated on a 7-point frequency scale (1 = never, 7 = several times an hour). A total score is calculated by summing all items, with higher scores indicating more severe agitation/sundowning. Change in CCMAI total score will be compared within participants across aromatherapy intervention phases.

SECONDARY OUTCOMES:
Change in sleep quality (Chinese Pittsburgh Sleep Quality Index, CPSQI) | Baseline and the end of each 2-week aromatherapy phase (up to 6 weeks)
  Sleep quality will be assessed using the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI). The CPSQI consists of 19 self- or proxy-rated items that generate seven component scores and a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality. For this study, the primary sleep outcome will be the global CPSQI score. Change in CPSQI global score will be compared within participants across the two aromatherapy phases.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Jy Wang, PhD, RN, Principal Investigator — National Cheng Kung University, College of Medicine, Department of Nursing
Locations (2):
- Taiwan (2):
  - Evergreen Senior Day Care Center, Kaohsiung, Taiwan
  - Kang Yu Day Care Center, Tainan, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared at this time. The dataset involves a small group of vulnerable older adults with dementia living in long-term care facilities, and the current IRB approval and informed consent do not include secondary data sharing. Only de-identified aggregate results will be reported in publications and presentations. IPD sharing may be considered in the future with additional ethics approval and appropriate data-sharing agreements to protect participant privacy.